CLINICAL TRIAL: NCT06833229
Title: Prospective Cohort Study Evaluating 18FDG PET-CT for the Early Prediction of the Efficacy of Immunotherapy Associated or Not With Chemotherapy in Patients With Locally Advanced or Metastatic Non-Small Cell Broncho-Pulmonary Carcinoma
Acronym: FDG Immun Comb
Status: Recruiting | Type: Observational
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/11; 2021-A00352-39 (Other: ANSM)
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung (NSCLC)
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: FDG-PET — PET scan are performed within 28 days before the start of immunotherapy, then at week 6 and week 12 of follow-up. Various metabolic parameters extracted from the standard PET image (ΔSUVmax, ΔTLG, appearance of new visceral lesion(s)), parametric (metabolic glucose rate (Ki), volume of distribution (VD)) and tumor response based on PERCIST criteria (adapted to immunotherapy) are assessed.

SUMMARY:
The hypothesis of this prospective observational pilot study of diagnostic diagnostic performance is that, for patients with NSCLC treated with immunotherapy associated or not with chemotherapy, certain metabolic biomarkers on 18FDG PET scans allow early identification of treatment response (or lack of response to treatment) and optimize prediction of tumor response compared with current standards.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years,
* Patients with histologically proven, metastatic or locally advanced NSCLC, with indication for immunotherapy (Nivolumab, pembrolizumab, atezolizumab, durvalumab, avelumab), in combination or not with chemotherapy molecules (carboplatin, cisplatin, pemetrexed, paclitaxel or nab-paclitaxel), validated by a Multidisciplinary Team and prescribed within the scope of their Marketed Authorization, whatever the line of treatment treatment line,
* ECOG 0 to 3,
* The patient's understanding of the protocol and the note of non-opposition, with oral agreement,
* Patient has not objected to the use of his or her data for medical research. research,
* Patient has social security coverage.

Exclusion Criteria:

* Age under 18,
* Contraindication to 18FDG PET-CT examinations: severe claustrophobia, unbalanced diabetes at the time of the first PET-CT scan (fasting capillary glucose ≥ 11 mmol),
* Hemoglobin less than 7 g/dL at inclusion. If the patient has a respiratory or or cardiovascular pathology, hemoglobin must not be less than 9.0 g/dL,
* Any participation in other biomedical studies involving the drug, medical devices or medical devices or imaging techniques is prohibited, with the exception of biomedical studies,
* Refusal to participate in the present study,
* Contraindication (e.g. hypersensitivity to the active substance or to one of the excipients of immunotherapy or chemotherapy treatments...).
* Vulnerable persons are defined in article L1121-5 to -8:

  * Pregnant women, parturients and nursing mothers, persons deprived of their liberty by judicial or administrative decision, persons hospitalized without consent under articles L. 3212-1 and L. 3213-1 who are not covered by the provisions of the provisions of article L. 1121-8,
  * and persons admitted to a health or social establishment for purposes other than research purposes,
  * adults who are the subject of a legal protection measure, or who are unable to exercise their non opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with locally advanced or metastatic NSCLC with an indication for immunotherapy combined with concomitant chemotherapy as standard treatment and managed at the Centre Antoine Lacassagne will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2028-05-27 (Estimated); Study Completion 2031-01-27 (Estimated)

PRIMARY OUTCOMES:
Metabolic criteria for PET imaging that can distinguish true tumor progression from pseudo-progression of inflammatory origin (leukocyte infiltrate) | 36 months
  Calculation of the area of the ROC curve and determination of the optimal threshold of different metabolic parameters extracted from the standard PET image (ΔSUVmax, ΔTLG, appearance of new visceral lesion(s)) and parametric PET image (metabolic glucose rate (Ki), volume of distribution (VD)) to distinguish lesions between true progression from inflammatory pseudoprogressions.

SECONDARY OUTCOMES:
Incidence of pseudo-progressions versus true tumor progressions at the first PET scan at 6 weeks. | 6 weeks
  Evaluation of the ratio between lesions with pseudo-inflammatory progression and those with true tumor progression (defined a posteriori on control PET-CT). A analysis per lesion and per patient. Two groups of patients will be compared: the group treated with immunotherapy alone and the group treated with a combination of immunotherapy and chemotherapy
Prognostic value of metabolic response PET-CT at 6 weeks and 12 weeks on overall survival at 12, 24 and 36 months | 36 months
  Overall survival at 12, 24 and 36 months as a function of changes in tumor metabolism on the first interim PET-CT scans (PERCIST and ΔSUV analysis). Overall survival: time from date of inclusion to date of death from any cause.
Use of supervised deep-learning algorithms (neural networks) to classify patients as immunotherapy responders or non-responders. | 6 months
  Non-responders will be defined as patients who discontinue immunotherapy within the first 6 months of treatment due to tumor progression. Responders will be defined by continuation of immunotherapy beyond 6 months of treatment.
Evaluation of overall survival of patients with oligometastatic progression with maintenance of immunotherapy and targeted irradiation of progressing lesions. | 36 months
  Overall survival at 24 months as a function of whether or not irradiation (as part of standard practices) of progressing lesions in patients with metastatic oligo-progression on 18FDG PET (between 1 and 3 progressive lesions).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine Lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided